CLINICAL TRIAL: NCT01931423
Title: The Influence of Placental Drainage of Management of the Third Stage of Labor:a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, M.D. Obstetric and Gynecology, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Aşıcıoğlu-06
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2013-11

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

ARMS (2):
- Drainage Group (Placebo Comparator): early placental drainage plus cord traction
  Interventions: Behavioral: Placental cord drainage
- Controlled Group (No Intervention): spontaneous removal placenta

INTERVENTIONS:
Behavioral: Placental cord drainage
  Arms: Drainage Group

SUMMARY:
To determine whether early placental drainage plus cord traction reduces the incidences of manual removal and blood loss, and to determine the risk factors associated with blood loss after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. greater than 37 gestational weeks
2. single pregnancy
3. vaginal delivery
4. estimated fetal weight 2500-4500 gr.

Exclusion Criteria:

1. PPROM
2. 37 or lower gestational week
3. multiple pregnancy
4. grand multiparıty (greater than 5)
5. coagulation defects (HELLP, ablation placenta, previa, pre-eclampsia)
6. a history of any bleeding during pregnancy
7. caesarean delivery or any uterine scar
8. a history of postpartum haemorrhage
9. hydramnios
10. known uterine anomalies
11. suspected abnormal placentation (accreta, increta, or percreta)
12. prepartum hemoglobin concentration less than 8 g/dL
13. history of anticoagulant drugs and prolongation of the first stage of labor longer than 15 hours

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 485 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
postpartum blood loss | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Osman Aşıcıoğlu, M.D., Principal Investigator — T.C.S.B. Şişli Etfal Research Hospital
Locations (1):
- Osman Aşıcıoğlu, Istanbul, ŞiŞLİ, Turkey (Türkiye)